CLINICAL TRIAL: NCT01396512
Title: Immunogenicity and Safety of a Single Dose of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV™) in Comparison With a Single Dose of SA14-14-2 Vaccine (CD.JEVAX™, Chengdu Institute of Biological Products, China) Administered in Healthy Toddlers in South-Korea
Brief Title: Study of a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV™) Compared to CD.JEVAX™ in Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JEC12; U1111-1117-7378 (Other: WHO)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-03

CONDITIONS: Japanese Encephalitis; Japanese Encephalitis Virus Disease
Keywords: Japanese Encephalitis; Japanese Encephalitis Virus Disease; IMOJEV™; CD.JEVAX™
MeSH Terms: conditions — Encephalitis, Japanese | interventions — SA-14-14-2 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMOJEV™ Vaccine Group (Experimental): Participants will receive a single dose of the Live attenuated Japanese encephalitis chimeric virus vaccine (IMOJEV™) on Day 0.
  Interventions: Biological: Live attenuated Japanese encephalitis chimeric virus vaccine
- CD.JEVAX ™ Vaccine Group (Active Comparator): Participants will receive a single dose of the Japanese encephalitis live attenuated vaccine (SA14 14 2 vaccine), CD.JEVAX™ on Day 0
  Interventions: Biological: Japanese encephalitis live attenuated vaccine (SA14 14 2 vaccine)

INTERVENTIONS:
Biological: Live attenuated Japanese encephalitis chimeric virus vaccine — 0.5 mL, Subcutaneous
  Other Names: IMOJEV™
  Arms: IMOJEV™ Vaccine Group
Biological: Japanese encephalitis live attenuated vaccine (SA14 14 2 vaccine) — 0.5 mL, Subcutaneous
  Other Names: CD.JEVAX™
  Arms: CD.JEVAX ™ Vaccine Group

SUMMARY:
The purpose of this study is to compare Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV™) with Japanese encephalitis live attenuated vaccine (SA14 14 2 vaccine [CD.JEVAX™]) after a single dose vaccination to support product registration.

Primary Objective:

* To demonstrate the non-inferiority of the antibody response 28 days after administration of one dose of IMOJEV™ compared to the antibody response 28 days after administration of one dose of the CD.JEVAX™ control vaccine.

Secondary Objectives:

* To describe the immune response to Japanese encephalitis (JE) in both vaccine groups using 50% plaque reduction neutralization assay (PRNT50) assays before and after a single dose of IMOJEV™ vaccine or a single dose of CD.JEVAX™ vaccine.
* To describe the safety of vaccination in all subjects up to 28 days and all serious adverse events up to 6-month after vaccination.

DETAILED DESCRIPTION:
All participants will receive a single dose of their assigned vaccination at Visit 1 (Day 0) and undergo immunogenicity assessment at Day 28 post-vaccination. Safety will be assessed from day of vaccination and up to 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 24 months on the day of inclusion
* In good general health, without significant medical history.
* Provision of informed consent form signed by at least one parent or other legally acceptable representative.
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Known systemic hypersensitivity to any of IMOJEV™ components or history of a life-threatening reaction to a vaccine containing any of the same substances and vaccination,known systemic hypersensitivity to CD.JEVAX® main components and the other components (including Gelatin, kanamycin, and gentamicin).
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of the immune response.
* Previous vaccination against flavivirus disease, including Japanese encephalitis (JE).
* Administration of any anti-viral within 2 months preceding Visit 01 and up to the 4 weeks following the trial vaccination.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination, except for pandemic influenza vaccination, which may be received at least two weeks before the study vaccines.
* Planned receipt of any vaccine from the inclusion up to the 4 weeks following the trial vaccination.
* History of central nervous system disorder or disease, including seizures.
* Planned receipt of any JE vaccine during the course of the study.
* History of flavivirus infection (confirmed either clinically, serologically or virologically).
* Administration of systemic corticosteroids for more than two consecutive weeks within the 4 weeks preceding vaccination.
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection 3 days before vaccination as well as the day of vaccination, according to Investigator judgment.
* Thrombocytopenia or bleeding disorder contraindicated for vaccination with same administration route, or receipt of anticoagulants in the 3 weeks preceding inclusion.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (6):
- South Korea (6):
  - Goyang
  - Incheon
  - Seongnam
  - Seoul
  - Suwon
  - Wŏnju

REFERENCES:
- [Derived] Kim DS, Houillon G, Jang GC, Cha SH, Choi SH, Lee J, Kim HM, Kim JH, Kang JH, Kim JH, Kim KH, Kim HS, Bang J, Naimi Z, Bosch-Castells V, Boaz M, Bouckenooghe A. A randomized study of the immunogenicity and safety of Japanese encephalitis chimeric virus vaccine (JE-CV) in comparison with SA14-14-2 vaccine in children in the Republic of Korea. Hum Vaccin Immunother. 2014;10(9):2656-63. doi: 10.4161/hv.29743. Epub 2014 Nov 6. PMID 25483480
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 12 July 2011 to 28 September 2012 at 10 clinic centers in South Korea.
Pre-assignment Details: A total of 274 participants who met all of the inclusion and none of the exclusion criteria were randomized and vaccinated in this study.
Groups:
- IMOJEV™ Vaccine Group: Participants age 12 to 24 months received one dose of IMOJEV™
- CD.JEVAX™ Vaccine Group: Participants age 12 to 24 months received one dose of CD.JEVAX™
Period: Overall Study
Arm/Group | IMOJEV™ Vaccine Group | CD.JEVAX™ Vaccine Group
Started | 137 | 137
Completed | 137 | 136
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMOJEV™ Vaccine Group | CD.JEVAX™ Vaccine Group | Total
Number analyzed (Participants) | 137 | 137 | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 137 | 137 | 274
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.0 (2.0) | 14.3 (2.2) | 14.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 57 | 115
  Male | 79 | 80 | 159
Region of Enrollment [Number; unit: Participants]
  South Korea | 137 | 137 | 274

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion to Japanese Encephalitis Chimeric Virus Following Vaccination With Either IMOJEV™ or CD.JEVAX™ Japanese Encephalitis Vaccine
Description: Immunogenicity assessed using a Japanese encephalitis chimeric virus (JE-CV) 50% Plaque Reduction Neutralization Test (PRNT50). Seroconversion was defined as the percentage of participants who developed neutralizing antibody titers above 10 (1/dil) when seronegative at baseline (<1/10) or who presented a ≥4-fold rise in their neutralizing antibody titers when seropositive (≥1/10) at baseline.
Time Frame: Day 28 post-vaccination
Population: Seroconversion to JE-CV was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | IMOJEV™ Vaccine Group | CD.JEVAX™ Vaccine Group
Number analyzed (Participants) | 119 | 117
Percentage of Participants | 100 | 99.1

2. Secondary Outcome: Geometric Mean Titers Against the Japanese Encephalitis Chimeric Virus Before And Following Vaccination With Either IMOJEV™ or CD.JEVAX™ Japanese Encephalitis Vaccine
Description: Geometric mean titers were assessed using a Japanese encephalitis chimeric virus (JE-CV) 50% Plaque Reduction Neutralization Test (PRNT50).
  JE-CV PRNT50 antibody titer >10 (1/dil, Day 0)
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers against the JE-CV was assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | IMOJEV™ Vaccine Group | CD.JEVAX™ Vaccine Group
Number analyzed (Participants) | 119 | 117
Titers
  JE-CV PRNT50 antibody titer (pre-vaccination) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  JE-CV PRNT50 antibody titer (post-vaccination) | 908 [656 to 1256] | 579 [427 to 784]

3. Secondary Outcome: Number of Participants With Seroprotection Against Japanese Encephalitis Chimeric Virus Before And Following Vaccination With Either IMOJEV™ or CD.JEVAX™ Japanese Encephalitis Vaccine
Description: Immunogenicity was assessed using a Japanese encephalitis chimeric virus (JE-CV) PRNT50 assay. Seroprotection was defined as the percentage of participants with a titer ≥10 (1/dil) at pre-vaccination and at Day 28 post-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection against JE-CV was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | IMOJEV™ Vaccine Group | CD.JEVAX™ Vaccine Group
Number analyzed (Participants) | 119 | 117
Participants
  JE-CV PRNT50 antibody titer ≥10 (1/dil, Day 0) | 0 | 0 [0 to 0]
  JE-CV PRNT50 antibody titer ≥10 (1/dil, Day 28) | 119 | 116 [0 to 0]

4. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Following Vaccination With Either IMOJEV™ or CD.JEVAX™ Japanese Encephalitis Vaccine
Description: Solicited injection site: Pain, Erythema, and Swelling; Solicited systemic reactions: Fever (Temperature), Vomiting, Crying Abnormal, Drowsiness, Appetite Loss, and Irritability. Grade 3 injection site: Pain - Cries when injected limb is moved or the movement of injected limb is reduced; Erythema and Swelling longest diameter ≥50 mm. Grade 3 systemic reactions: Fever >39.5°C; Vomiting ≥6 episodes per 24 hours or requiring parenteral hydration; Crying Abnormal - >3 hours; Drowsiness - sleeping most of the time or difficult to wake; Appetite Loss - refuses ≥3 feeds or most feeds; Irritability - inconsolable.
Time Frame: Day 0 up to Day 14 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | IMOJEV™ Vaccine Group | CD.JEVAX™ Vaccine Group
Number analyzed (Participants) | 137 | 137
Participants
  Injection site Pain (N = 137, 137) | 35 | 38 [0 to 0]
  Grade 3 Injection site Pain (N = 137, 137) | 0 | 1 [0 to 0]
  Injection site Erythema (N = 137, 137) | 23 | 33 [0 to 0]
  Grade 3 Injection site Erythema (N = 137, 137) | 0 | 0 [0 to 0]
  Injection site Swelling (N = 137, 137) | 6 | 10 [0 to 0]
  Grade 3 Injection site Swelling (N = 137, 137) | 0 | 0 [0 to 0]
  Fever (N = 134, 136) | 33 | 34 [0 to 0]
  Grade 3 Fever (N = 134, 136) | 1 | 1 [0 to 0]
  Vomiting (N = 137, 137) | 9 | 14 [0 to 0]
  Grade 3 Vomiting (N = 137, 137) | 1 | 2 [0 to 0]
  Crying Abnormal (N = 137, 137) | 27 | 35 [0 to 0]
  Grade 3 Crying Abnormal (N = 137, 137) | 2 | 3 [0 to 0]
  Drowsiness (N = 137, 137) | 23 | 33 [0 to 0]
  Grade 3 Drowsiness (N = 137, 137) | 0 | 1 [0 to 0]
  Appetite Loss (N = 137, 137) | 38 | 40 [0 to 0]
  Grade 3 Appetite Loss (N = 137, 137) | 4 | 1 [0 to 0]
  Irritability (N = 137, 137) | 31 | 36 [0 to 0]
  Grade 3 Irritability (N = 137, 137) | 1 | 5 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination.
Arm/Group | IMOJEV™ Vaccine Group | CD.JEVAX™ Vaccine Group
Serious Adverse Events (participants affected / at risk) | 17/137 | 18/137
Other Adverse Events (participants affected / at risk) | 74/137 | 69/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMOJEV™ Vaccine Group (N=137) | CD.JEVAX™ Vaccine Group (N=137)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (2)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Hand foot and mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 1 (1) | 0 (0)
Lymph node abscess (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Kawasaki's disease (Nervous system disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IMOJEV™ Vaccine Group (N=137) | CD.JEVAX™ Vaccine Group (N=137)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 3 (3)
Pyrexia (General disorders) | 8 (8) | 9 (9)
Bronchitis (Infections and infestations) | 9 (9) | 6 (7)
Gastroenteritis (Infections and infestations) | 4 (4) | 7 (8)
Nasopharyngitis (Infections and infestations) | 42 (54) | 38 (44)
Otitis media (Infections and infestations) | 6 (7) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 11 (13) | 4 (5)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 7 (8)
Injection site Pain (General disorders) | 35 (35) | 38 (38)
Injection site Erythema (General disorders) | 23 (23) | 33 (33)
Injection site Swelling (General disorders) | 6 (6) | 10 (10)
Fever (General disorders) | 33/134 (33) | 34/136 (34)
Vomiting (Gastrointestinal disorders) | 9 (9) | 14 (14)
Crying Abnormal (Psychiatric disorders) | 27 (27) | 35 (35)
Drowsiness (Nervous system disorders) | 23 (23) | 33 (33)
Appetite Loss (Metabolism and nutrition disorders) | 38 (38) | 40 (40)
Irritability (Psychiatric disorders) | 31 (31) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.